CLINICAL TRIAL: NCT03926572
Title: Pronostic Study of Biomarkers in Acute Decompensation of Pulmonary Hypertension
Brief Title: Acute Decompensation of Pulmonary Hypertension
Acronym: PROPULS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP180273
Record Dates: First submitted 2019-04-15; First posted 2019-04-24 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-09

CONDITIONS: Hypertension, Pulmonary; Biomarkers
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Intervention Model Description: patients admitted for acute decompensation of pulmonary arterial hypertension or postembolic pulmonary hypertension with samples of blood samples taken at admission, days 3 and 7 in the context of this clinical study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Pulmonary arterial hypertension (Other): Pulmonary arterial hypertension or non-operable chronic thromboembolic pulmonary hypertension established by right cardiac catheterization prior to inclusion in the study
  Interventions: Other: A biobank will be created from blood samples taken at admission, days 3 and days 7

INTERVENTIONS:
Other: A biobank will be created from blood samples taken at admission, days 3 and days 7 — A biobank will be created from the blood samples taken on admission, days 3 and 7 of admission. The prognostic value of the preselected biomarkers will be analyzed and a proteomic analysis will be performed to identify new biomarkers. The prognostic value of these new biological parameters will be compared to the usual surveillance parameters that will be collected during the follow-up (clinical, echocardiographic and hemodynamic parameters)

SUMMARY:
The main objective of this study is to analyze the survival of a cohort of patients admitted for acute decompensation of pulmonary arterial hypertension or postembolic pulmonary hypertension and to establish the prognostic value of biomarkers.

DETAILED DESCRIPTION:
It is planned to include 150 patients over a two-year period. The primary endpoint is a composite endpoint including death, circulatory assistance or emergency transplantation within 90 days following admission to intensive care unit. Patients will be treated according to the usual practice. A biobank will be created from blood samples taken at admission, days 3 and days 7. Prognostic value of pre-selected biomarkers will be analyzed and a proteomic analysis will be performed in order to identify new biomarkers. The prognostic value of these new biological parameters will be compared to the usual monitoring parameters that will be collected during follow-up (clinical, echocardiographic and haemodynamic parameters). In a second step, it will establish, using a dynamic model, the best combinations of parameters allowing to best assessment of prognosis of patients suffering from PH and hospitalized for acute right ventricular failure.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over 18 years
* Diagnosis of Pulmonary arterial hypertension or non-operable chronic thromboembolic pulmonary hypertension established by right cardiac catheterization prior to inclusion in the study
* Patients admitted in intensive care unit for acute decompensation of pulmonary hypertension requiring intravenous diuretic therapy ± use of inotropes or vasopressors.
* Patients must have given their written informed consent to participate in the study after having received adequate previous information and prior to any study-specific procedures

Exclusion Criteria:

* Patients with post-capillary pulmonary hypertension
* Patients with pulmonary hypertension associated with chronic respiratory disease
* Patients with pulmonary hypertension with unclear/or multifactorial mechanisms
* Patients with operable chronic thromboembolic pulmonary hypertension
* Shock due to another cause than acute decompensation of pulmonary hypertension
* Pregnant women, or breast feeding women
* Adult protected person
* Person deprived of liberty
* Person admitted without consent
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
time to death, circulatory assistance or emergency transplantation within 90 days following admission to intensive care unit | 90 days
  The primary endpoint is a composite endpoint including death, circulatory assistance or emergency transplantation within 90 days following admission to intensive care unit

SECONDARY OUTCOMES:
Survival time without graft or circulatory assistance | 1 month
  Survival without transplantation or circulatory assitance at 1 month
Survival time without transplantation or circulatory assitance | 12 months
  Survival ithout transplantation or circulatory assitance at 12 month

CONTACTS AND LOCATIONS:
Overall Officials: SAVALE Laurent, MD, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- SAVALE Laurent, Le Kremlin-Bicêtre, France